CLINICAL TRIAL: NCT06273670
Title: Regular Six Weeks Versus Earlier Postpartum Initiation of Long-acting Reversible Contraceptives: Knowledge Attitude and Practice Study (KAP)
Brief Title: Postpartum Initiation of Long-acting Reversible Contraceptives: Knowledge Attitude and Practice Study (KAP)
Acronym: KAP
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Mahmoud M. Khalil, Doctor, Assiut University
Other Study IDs: 04-2023-200279
Record Dates: First submitted 2023-07-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Contraception
Keywords: Postpartum contraception; LARC; KAP
MeSH Terms: interventions — Mass Screening; Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Service providers: General practitioners, specialists, nurses, and social workers.
  Interventions: Other: screening and data collection
- Clients: All clients who were attending family planning centers in public health facilities at the study period will be included if they have had a postpartum LARC method (Copper IUD, Progestin-releasing IUS or Subdermal implant) or willing to use it in the first year after delivery.
  Interventions: Other: screening and data collection

INTERVENTIONS:
Other: screening and data collection — Structured questionnaire prepared in English and translated to local language (Arabic). The questionnaire is then linguistically validated by two forwards translations and one backward translation. Data was collected by the investigators who were not participating in the study.
  Personal or telephone interview will be conducted with clients and service providers conducted to collect the data.

SUMMARY:
Comparing Knowledge, attitude and Practice of clients and service providers about the regular (6 weeks) versus earlier initiation of LARC, through a structured questionnaire prepared in English and translated to local language i.e. Arabic.

DETAILED DESCRIPTION:
Family planning is a behavior that allows individuals and couples to anticipate and attain their desired number of children, at the spacing and timing of their births. It is achieved through the use of contraceptive methods and treatment of involuntary infertility.

Postpartum family planning is the prevention of unintended and closely spaced pregnancies during the first 12 months following childbirth. Short interval pregnancies are associated with increased maternal morbidities such as anemia, bleeding disorders, premature rupture of membranes, puerperal endometritis and mortality .

Postpartum family planning (PPFP) has long been recognized as an important component of maternal health care. Through birth spacing and prevention of high-risk and unwanted pregnancies, PPFP helps women who have recently delivered to avoid exposure to the risks of maternal death. Likewise, the importance of the interplay between maternal health services and use of contraception in the postpartum period has been recognized for decades.

Globally, more than 90 percent of women during the first year postpartum want to either delay or avoid future pregnancies . An increase in contraceptive use during the postpartum period should substantially reduce rates of maternal and infant mortality by preventing unplanned and unwanted pregnancies and by spacing new pregnancies at least two years after the previous birth .

ELIGIBILITY:
Inclusion Criteria:

Client's group All clients who were attending family planning centers in public health facilities at the study period if they have had a postpartum LARC method (Copper IUD, Progestin-releasing IUS, Subdermal implant) or willing to use it in the first year after delivery.

Service provider group:

All service providers who are working in primary health care units & hospitals, including general practitioners, ob/gyn. specialists, nurses, and social workers.

Exclusion Criteria:

* Clients and service providers who refused to participate in the study
* Clients who are currently using or willing to use a method other than LARC

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Client's group:
  All females visiting family planning centers in public health facilities who delivered within a year and receiving a LARC method or willing are asked to volunteer.
  Service provider group:
  All service providers who are working in primary health care units & hospitals, including general practitioners, ob/gyn. specialists, nurses, and social workers are asked to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Clients' knowledge | Immediately. The outcome is provided in the questionnaire which is completed once by the client
  The percentage of clients who have good knowledge that LARC can be initiated early after delivery

SECONDARY OUTCOMES:
Clients' attitude | Immediately. The outcome is provided in the questionnaire which is completed once by the client
  The percentage of clients who have positive attitude towards early initiation of LARC after delivery
Clients' practice | Immediately. The outcome is provided in the questionnaire which is completed once by the client
  The percentage of clients who had previously or lately initiated any LARC early after delivery
Providers' knowledge | Immediately. The outcome is provided in the questionnaire which is completed once by the client
  The percentage of providers who have good knowledge that LARC can be initiated early after delivery
Providers' attitude | Immediately. The outcome is provided in the questionnaire which is completed once by the client
  The percentage of providers who have positive attitude towards early initiation of LARC after delivery
Providers' practice | Immediately. The outcome is provided in the questionnaire which is completed once by the client
  The percentage of providers who had previously or lately initiated any LARC for women early after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali Abdelaleem, Doctorate, Study Chair — Obstetrics and gynecology department, Assiut University; Karim abdelhameed, Doctorate, Study Chair — Obstetrics and gynecology department, Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Committee Opinion No. 642: Increasing Access to Contraceptive Implants and Intrauterine Devices to Reduce Unintended Pregnancy. Obstet Gynecol. 2015 Oct;126(4):e44-e48. doi: 10.1097/AOG.0000000000001106. PMID 26393458
- [Background] Washington CI, Jamshidi R, Thung SF, Nayeri UA, Caughey AB, Werner EF. Timing of postpartum intrauterine device placement: a cost-effectiveness analysis. Fertil Steril. 2015 Jan;103(1):131-7. doi: 10.1016/j.fertnstert.2014.09.032. Epub 2014 Oct 25. PMID 25439838
- [Result] Conde-Agudelo A, Belizan JM. Maternal morbidity and mortality associated with interpregnancy interval: cross sectional study. BMJ. 2000 Nov 18;321(7271):1255-9. doi: 10.1136/bmj.321.7271.1255. PMID 11082085